CLINICAL TRIAL: NCT05805592
Title: The Effect of Screen to Move Program (STEP) on Screen Use Time and Physical Activity in Preschool Children
Brief Title: The Effect of Screen to Move Program in Preschool Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tuba Bay Kula, Principal Investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19092293
Record Dates: First submitted 2023-03-05; First posted 2023-04-10 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Physical Activity; Screen Time; Child, Preschool
Keywords: Physical Activity; Screen time; Pre-school child
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This study is a parallel group randomized controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): It is planned as 6 sessions, 1 session per week for children and parents. The program will be introduced to children and parents under the call with "Screen-to-Move-Program (STEP)". The symbol of the program has been created and this symbol will be hung on the classroom door. Sessions for children include story, picture, video demonstration and active playing activities. A more clear, simple and understandable language will be used for children, and reinforcements will be used. For parents; There will be 6 training sessions in the form of presentations. At the same time as the children's activities, information notes will be sent to the parents outlining the expectations. Before the intervention, after the intervention and in the 3rd month, children's screen use time, daily physical activity time, sleep time, parents' knowledge, behavior, attitude and self-efficacy about their children's screen use time will be evaluated.
  Interventions: Behavioral: Screen-to-Move-Program (STEP)
- Control Group (No Intervention): Screen use time, daily physical activity time, sleep time, parents' knowledge, behavior, attitude and self-efficacy about children's screen use time will be evaluated simultaneously from the control group with the intervention group. After the 3rd month follow-up test, the STEP will be applied to the children and parents in the control group.

INTERVENTIONS:
Behavioral: Screen-to-Move-Program (STEP) — It is planned as 6 sessions, 1 session per week for children and parents. The program will be introduced to children and parents under the call with "Screen-to-Move-Program (STEP)".
  Arms: Intervention Group

SUMMARY:
The aim of this study is to determine the effect of the developed program on screen usage time and physical activity for pre-school children.

DETAILED DESCRIPTION:
The "Screen-to-Move-Program" (STEP), developed on the basis of Social Cognitive Theory (SCT), is aimed to reduce screen usage time and increase physical activity in pre-school children. In this study, it was aimed to increase children's physical activity and decrease screen usage times with a 6 session intervention program based on SCT, which includes children and parents. The effectiveness of the program will be evaluated with the pre-test, post-test and 3rd month follow-up test.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 36-60 months and their parents.
2. Children without any physical and mantel disability

Exclusion Criteria:

1.The data of parents who fill in the data collection forms incompletely will be excluded from the analysis

Ages: 36 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Decreasing screen time of children in the experimental group | Change in screen usage time within 3 months
  Children's screen usage time will be evaluated with questions. "How long (…hours…..minutes) on average did your child use any device with an electronic screen, such as a smartphone, tablet, video game, or watch television, movies, video games in a day?". Daily screen usage time will be evaluated in minutes. A maximum of 60 minutes of screen time is recommended for pre-school children (World Health Organization, 2019).
Increasing physical activity level of children in the experimental group | Change in physical activity level within 3 months
  Children's physical activity levels; Item 1: "How long is your child active on average in a day? (e.g. walking slowly, making the bed etc.)" and Item 2:"How long does your child do physical activity in a day, on average, until he is out of breath?" (walking fast, cycling, running, playing ball games, swimming, dancing, etc.) will be evaluated based on parent self-report. The total daily (Item1 + Item2) physical activity time will be evaluated in minutes. A minimum of 180 minutes of physical activity is recommended for pre-school children (World Health Organization, 2019).
Increasing number of steps for the children in the experimental group | Change in number of steps within 3 months
  Pre-school children's daily step count will be measured with the OMRON HJ-109-E pedometer. In our study, the number of steps for children aged 3-5 will be evaluated as 11,500 steps, which is stated to correspond to the 180 minutes physical activity target recommended by the World Health Organization for children aged 3-5 (De Craemer et al., 2015; World Health Organization, 2019).

SECONDARY OUTCOMES:
Increasing knowledge score of parents in the experimental group | Change in knowledge score of parents within 3 months
  The information form was created by researchers in line with the literature (World Health Organization, 2019). The form contains information about the PA, screen usage time and sleep duration of the children of parents who have children between the ages of 2-5 and consists of 14 questions. For each item, the correct option is scored as 1, and the incorrect and I don't know option is scored as 0. The total score obtained by collecting the items varies between 0-14 points. A high score indicates a high level of knowledge.
Increase in the attitude score of the parents in the experimental group | Change in parents' attitudes within 3 months
  Parents' attitudes towards their children's screen time were evaluated with an eight-item questionnaire developed by Zimmerman et al. in 2007. The questionnaire is in a five-point Likert type, ranging from strongly agree (1) to strongly disagree (5). High scores on the survey reflect more positive attitudes. The questionnaire has been used in many studies before and has a high reliability with the cronbach alpha value of .84 (Carson & Janssen, 2012; Mansor et al., 2021; Raj et al., 2022).
Increasing self-efficacy score of parents in the experimental group | Change in self-efficacy score of parents within 3 months
  Self-efficacy will be measured separately to reduce screen time and increase physical activity. Parents' self-efficacy in reducing their children's screen time: "How confident are you that you can say no to your child's request to participate in screen time (TV/computer/tablet/video games)?" It will be assessed on a 5-point scale ranging from 'not at all sure' to 'very sure' (Carson & Janssen, 2012). The parent's self-efficacy in influencing the child's physical activity reflects the parent's level of confidence in situations related to the child's physical activity. The questionnaire developed in 2010 has a single factor structure and high reliability (α= 0.88). The eight-question survey (For example: How confident are you that your child will do physical activity even if you do not have much time) is a five-point Likert type ranging from I do not trust myself (1) to I am very confident (5). High scores on the questionnaire reflect higher self-efficacy (Smith et al., 2010).

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Ergun, Prof, Study Chair — Marmara University; Tuba Bay Kula, MSc, RN, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carson V, Janssen I. Associations between factors within the home setting and screen time among children aged 0-5 years: a cross-sectional study. BMC Public Health. 2012 Jul 23;12:539. doi: 10.1186/1471-2458-12-539. PMID 22823887
- [Result] De Craemer M, De Decker E, De Bourdeaudhuij I, Verloigne M, Manios Y, Cardon G. The translation of preschoolers' physical activity guidelines into a daily step count target. J Sports Sci. 2015;33(10):1051-7. doi: 10.1080/02640414.2014.981850. Epub 2014 Dec 18. PMID 25524541
- [Result] Mansor E, Ahmad N, Raj D, Mohd Zulkefli NA, Mohd Shariff Z. Predictors of Parental Barriers to Reduce Excessive Child Screen Time Among Parents of Under-Five Children in Selangor, Malaysia: Cross-sectional Study. J Med Internet Res. 2021 Apr 13;23(4):e25219. doi: 10.2196/25219. PMID 33847590
- [Result] Raj D, Mohd Zulkefli N, Mohd Shariff Z, Ahmad N. Determinants of Excessive Screen Time among Children under Five Years Old in Selangor, Malaysia: A Cross-Sectional Study. Int J Environ Res Public Health. 2022 Mar 17;19(6):3560. doi: 10.3390/ijerph19063560. PMID 35329247
- [Result] Smith BJ, Grunseit A, Hardy LL, King L, Wolfenden L, Milat A. Parental influences on child physical activity and screen viewing time: a population based study. BMC Public Health. 2010 Oct 8;10:593. doi: 10.1186/1471-2458-10-593. PMID 20929587
- [Result] Zimmerman FJ, Christakis DA, Meltzoff AN. Television and DVD/video viewing in children younger than 2 years. Arch Pediatr Adolesc Med. 2007 May;161(5):473-9. doi: 10.1001/archpedi.161.5.473. PMID 17485624
- [Result] Guidelines on Physical Activity, Sedentary Behaviour and Sleep for Children under 5 Years of Age. Geneva: World Health Organization; 2019. Available from http://www.ncbi.nlm.nih.gov/books/NBK541170/ PMID 31091057